CLINICAL TRIAL: NCT03263273
Title: A Multicenter, Randomized, Double-Blind, Parallel Group, Vehicle-Controlled Study to Evaluate the Safety and Efficacy of 1% and 3% Topical MIinocycline Gel (HY01) in Patients With Papulopustular Rosacea
Brief Title: Study to Evaluate the Safety and Efficacy of Topical Minocycline Gel in Patients With Papulopustular Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hovione Scientia Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HY01-003
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Rosacea; Papulopustular Rosacea
Keywords: Minocycline; Topical; Tetracycline; Doxycycline; Rosacea; Skin Disease; Anti-Bacterial Agent; Anti-Inflammatory Agent
MeSH Terms: conditions — Rosacea; cyclopia sequence; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Topical Vehicle Gel (Placebo Comparator): Topical administration of vehicle gel. Regimen: Apply once daily, at bedtime to the face
  Interventions: Other: Topical Vehicle Gel
- 1% Topical Minocycline Gel (Active Comparator): Topical administration of 1% Topical Minocycline Gel. Regimen: Apply once daily, at bedtime to the face
  Interventions: Drug: 1% Topical Minocycline Gel
- 3% Topical Minocycline Gel (Active Comparator): Topical administration of 3% Topical Minocycline Gel. Regimen: Apply once daily, at bedtime to the face
  Interventions: Drug: 3% Topical Minocycline Gel

INTERVENTIONS:
Drug: 1% Topical Minocycline Gel — Treating Papulopustular Rosacea while monitoring for safety and efficacy of the active intervention
  Other Names: HY01 Topical Gel, 1%
  Arms: 1% Topical Minocycline Gel
Drug: 3% Topical Minocycline Gel — Treating Papulopustular Rosacea while monitoring for safety and efficacy of the active intervention
  Other Names: HY01 Topical Gel, 3%
  Arms: 3% Topical Minocycline Gel
Other: Topical Vehicle Gel — Treating Papulopustular Rosacea while monitoring for safety and efficacy of the vehicle intervention
  Other Names: HY01 Topical Gel, 0%
  Arms: Topical Vehicle Gel

SUMMARY:
To evaluate the efficacy of once-daily application of 1% and 3% HY01 Topical Gel, as assessed by the change in inflammatory lesion count from baseline over the 12-week treatment period in patients with moderate-to-severe papulopustular rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who had provided written informed consent to participate in the study.
* Male or non-pregnant female aged ≥ 18 years with a clinical diagnosis of moderate to severe facial rosacea, defined as the presence of: i. At least twelve and not more than forty inflammatory facial lesions (i.e., papules/pustules), AND ii. Subjects with a grade 3 or 4 on the 5-point Investigators Global Assessment (IGA) scale, AND iii. Persistent facial erythema (scored as at least mild on Erythema Severity Scale), AND iv. Facial telangiectasia (scored as at least mild on Telangiectasia Severity Scale.
* Subject willing to minimize external factors that might trigger rosacea flare-ups as recommended per protocol and patient instructional guide (e.g., spicy foods, thermally hot foods and drinks, hot environments, prolonged sun exposure, strong winds and alcoholic beverages).
* Non-nursing, female subjects of child bearing potential, who are using an acceptable form of birth control: total abstinence, oral (birth control pills), intravaginal: (e.g. NuvaRing®), implantable (e.g. Norplant®), injectable (e.g. Depo-Provera®) or transdermal (e.g. Ortho Evra®) contraception; intrauterine device (IUD); double-barrier (diaphragm or condom with spermicidal gel or foam); for two months prior to study enrollment or a vasectomized partner. All female subjects of child bearing potential must have undergone an in-office urine pregnancy test, with a negative result, prior to being randomized to receive study drug. In addition, women of childbearing potential must have agreed to a have urine pregnancy test at Day 42 and at the end of the study (Day 84). Females not of childbearing potential due to menopause must have been postmenopausal for at least one year. Male subjects must be willing to not attempt to conceive a child during the participation in the study. Females utilizing oral contraception must be willing to utilize an appropriate secondary form of contraception during the study.
* Subjects who use the same brand of soap, make-up, hair products, or shaving lotion/foam/cream/gel for a period of at least four weeks prior to the Baseline Visit and agree not to change these product brand/types during the study, with the exception of using the study approved cleanser and moisturizer with sunscreen provided by the sponsor.
* Male subjects who are willing to shave, if applicable, at approximately the same time every day.
* Subjects who are willing to refrain from sunbathing, using sun tanning booths/beds, or excessive exposure to the sun for the duration of the study.

Exclusion Criteria:

* Presence of any skin condition on the face that would interfere with the diagnosis or assessment of rosacea as determined by the Investigator.
* Excessive facial hair (e.g. beards, sideburns, moustaches, etc.) that would interfere with diagnosis or assessment of rosacea. Patients also must not grow excess facial hair during the study (i.e. they need to be free of excess facial hair for follow-up visits).
* History of hypersensitivity or allergy to minocycline, any other tetracycline or any other component of the formulation, or known reactions to cleansers, including Ponds Cold Cream, and moisturizer with sunscreen.
* Subjects using, or planning use of concomitant treatments within 30 days prior to Baseline visit (e.g., facial or chemical peels, dermal fillers, acne surgery, intralesional steroids, spironolactone, debridement, cryotherapy, dermabrasion, X-ray, IPL, laser therapy or UV therapy).
* Use within 6 months prior to baseline of oral retinoids (e.g. isotretinoin, acitretin) or therapeutic vitamin A supplements of greater than 10,000 International Units/day (multivitamins are allowed).
* Subjects using estrogens or progestin agents (e.g., Gynogen, Valergen, Depo-Testadiol, Depogen, birth control pills), for less than 2 months prior to the Baseline Visit. (Subjects using estrogens for 2 months or more are not excluded unless the subject expected to change dose, drug, or discontinue estrogen use during the study).
* Use within 2 month prior to the Baseline Visit of 1) topical retinoids to the face, 2) systemic antibiotics known to have an impact on the severity of facial rosacea (e.g., containing tetracycline and its derivatives, erythromycin and its derivatives, sulfamethoxazole, or trimethoprim, metronidazole), or 3) systemic corticosteroids.
* Use within 2 months prior to the Baseline Visit of 1) topical corticosteroids, 2) topical antibiotics or 3) topical medications for rosacea (e.g., metronidazole, azelaic acid, erythromycin, ivermectin, sulfur based topical products).
* Subjects with rhinophyma, dense telangiectasia, or plaque-like facial edema, more than 5 nodules or sinus tracts.
* Ocular rosacea (e.g., conjunctivitis, blepharitis, or keratitis) of sufficient severity to require topical or systemic antibiotics.
* Subjects with underlying diseases or other dermatological conditions, such as; atopic dermatitis, perioral dermatitis, or seborrheic dermatitis, which required the use of interfering topical or systemic therapy or may have interfered with the rosacea diagnosis.
* Subjects using an investigational drug or participating in an investigational study within 30 days of the Baseline Visit. Use of an investigational drug and/or participation in another investigational study prohibited during this study.
* Subjects who currently abuse alcohol or drugs or who have a history of chronic alcohol or drug abuse with in the past year.
* Medical history of immunodeficiency or other significant ongoing medical condition or disease as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Lesion Count | 12 weeks
  Evaluate the efficacy of once-daily application of 1% and 3% HY01 Topical Gel, as assessed by the change in inflammatory lesion count from baseline in patients with moderate-to-severe papulopustular rosacea

SECONDARY OUTCOMES:
Investigator's Global Assessment (IGA) Score | 12 weeks
  Evaluate the efficacy of once-daily application of 1% and 3% HY01 Topical Gel, in improving the Investigator's Global Assessment (IGA) scores from baseline over the 12-week treatment period in patients with moderate-to-severe papulopustular rosacea as defined as either a 2 point improvement from baseline or an improvement to "clear" or "almost clear" on the IGA

CONTACTS AND LOCATIONS:
Overall Officials: Sunil S Dhawan, MD, Principal Investigator — Center for Dermatology Clinical Research, Inc.
Locations (23):
- United States (23):
  - Clinical Site - 15, Bryant, Arkansas
  - Clinical Site - 20, Rogers, Arkansas
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Clinical Site - 19, Santa Monica, California
  - Clinical Site - 5, Tampa, Florida
  - Clinical Site - 16, Boise, Idaho
  - Clinical Site - 22, Boston, Massachusetts
  - Clinical Site - 23, Watertown, Massachusetts
  - Clinical Site - 14, Clinton Township, Michigan
  - Clinical Site - 6, Fridley, Minnesota
  - Clinical Site - 12, Omaha, Nebraska
  - Clinical Site - 21, Berlin, New Jersey
  - Clinical Site - 13, New York, New York
  - Clinical Site - 2, New York, New York
  - Clinical Site - 4, High Point, North Carolina
  - Clinical Site - 17, Portland, Oregon
  - Clinical Site - 11, Fort Washington, Pennsylvania
  - Clinical Site - 8, Goodlettsville, Tennessee
  - Clinical Site - 7, Pflugerville, Texas
  - Clinical Site - 18, San Antonio, Texas
  - Clinical Site - 3, San Antonio, Texas
  - Clinical Site - 9, San Antonio, Texas
  - Clinical Site - 10, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No